CLINICAL TRIAL: NCT02044900
Title: Polysomnography and Heart Rate Indexes in Obstructive Sleep Apnea
Status: Completed | Type: Observational
Sponsor: Ovidiu Constantin Baltatu (Other)
Responsible Party: Sponsor-Investigator, Ovidiu Constantin Baltatu, Professor, Universidade Camilo Castelo Branco
Organization: Universidade Camilo Castelo Branco (Other)
Other Study IDs: BR-001-SJC; 01328712.0.0000.5244 (Other: COMISSÃO NACIONAL DE ÉTICA EM PESQUISA - CONEP)
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; polysomnography; heart rate variability; mathematical biomarker
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the diagnostic accuracy of polysomnography indexes for diagnosis of sleep apnea in human subjects obstructive sleep apnea (OSA). This includes evaluation of polysomnography indexes (AHI; AI, arousal index; ODI, oxygen desaturation index) and heart rate variability (HRV) indexes.

DETAILED DESCRIPTION:
This is a cross-sectional study collecting data from patients from the Sleep Institute of Itaperuna, Rio de Janeiro, Brazil. Polysomnography (PSG) monitoring and diagnosis was in accordance with American Society of Sleep Medicine (ASSM) standards. Standard baseline polysomnography is performed using a computerised system. The following extracted signals are measured: 2 electroencephalogram channels (O1-A2, O2-A1, C3-A2, C4-A1), 2 electrooculogram channels, electromyography (EMG, bilateral anterior tibialis), pulse oximetry (arterial oxygen saturation), nasal-oral airflow (thermistors), and electrocardiogram (ECG derivation DII). The polysomnograms are scored according to the criteria of Rechtschaffen and Kales.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of obstructive sleep apnea with an apnea-hypopnea index (AHI) > 5.

Exclusion Criteria:

* Subjects with a history or clinical examination suggestive of neuromuscular disease, hypertension or any surgical treatment were not considered in the study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Polysomnography indexes | one night
  Polysomnography indexes and full-length sleep ECG recordings are extracted from polysomnogram measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Ovidiu C Baltatu, MD PhD, Study Chair — Camilo Castelo Branco University (UNICASTELO)
Locations (1):
- Sleep Institute of Itaperuna, Itaperuna, Rio de Janeiro, Brazil